CLINICAL TRIAL: NCT03894657
Title: Validation of Respiratory Epithelial Functional Assessment to Predict Clinical Efficacy of Orkambi®. Pathway to Personalized Therapy in Cystic Fibrosis
Brief Title: Validation of Respiratory Epithelial Functional Assessment to Predict Clinical Efficacy of Orkambi®.
Acronym: PREDICT-CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P170907J; 2018-002624-16 (EudraCT Number)
Record Dates: First submitted 2019-02-12; First posted 2019-03-28 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Cystic Fibrosis; Homozygous F508del Mutation
Keywords: CYSTIC FIBROSIS; ORKAMBI
MeSH Terms: conditions — Cystic Fibrosis | interventions — Blood Specimen Collection; lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Nasal brushing — Nasal scrapping at visit V0
Other: Sputum sample — Visit V0 : 1 Aliquot for Sputum biobank
  Visit V1 : 2 Aliquots
  * for Sputum biobank
  * for pharmacokinetic (PK) study
  Visit V2 : 2 Aliquots
  * for Sputum biobank
  * for pharmacokinetic (PK) study
Other: blood sample — Visit V0 : Additional 14 mL
  * 5 mL in ethylenediaminetetraacetic acid (EDTA) tube for DNA Analysis
  * 3 mL in Dry tube for Serum biobank
  * 6 mL in acid citrate dextrose (ACD) tube for peripheral blood mononuclear cell (PBMC) biobank
  Visit V1 : Additional 9 mL
  * 2x3 mL in dry tube for pharmacokinetic (PK) study
  * 3 mL in Dry tube for Serum biobank
  Visit V2 : Additional 6 mL
  * 3 mL in dry tube for pharmacokinetic (PK) study
  * 3 mL in Dry tube for Serum biobank
Drug: Orkambi — Study the predictive value for improvement of the respiratory function after 24 weeks of Orkambi treatment.
  Orkambi treatment is part of usual care.

SUMMARY:
The purpose of the study is to investigate whether the correction of CFTR function by Lumacaftor/Ivacaftor in a patient-derived primary nasal cell model is a surrogate biomarker for respiratory improvement in Orkambi® treated patients.

DETAILED DESCRIPTION:
Orkambi® is a combination of Ivacaftor (a CFTR channel potentiator) and Lumacaftor (a corrector partially rescuing the traffic of mutated CFTR). This treatment is now marketed in France for patients homozygotes for the mutation p.Phe508del, aged 12 and above. Systematic use of this product is a concern due to the lack of predictive markers of efficacy, the highly variable respiratory improvement in patients and potential serious side effects.

The purpose of this study is to investigate the predictive value for improvement of the respiratory function after 24 weeks of Orkambi treatment of an in vitro test. This test quantifies the correction of CFTR activity as assessed by the change of cyclic AMP (cAMP) dependant chloride (Cl-) secretion in patient derived Human Nasal Epithelial (HNE) derived primary culture after Lumacaftor/Ivacaftor 48 hours incubation.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous F508del patient aged 5 years or older
* Patient with an indication for Orkambi® treatment according to the marketing authorization application
* Patient never received Orkambi® in the past
* Patient able to perform FEV1
* Signed Informed consent form by the patient (if aged ≥ 18 years), or by parents / legal guardian and patient's agreement (if aged < 18 years) Patient affiliated to the health insurance system

Exclusion Criteria:

* Homozygous F508del patients who do not meet the treatment indications according to the marketing authorization application
* Patients refusing Orkambi®
* CF patients not homozygous for the p.Phe508del mutation
* Active smoker
* Severe nasal mucosa disrepair
* Contraindications to xylocaine anesthesia,
* Participation with another interventional study with drug

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Percentage of FEV1 | Baseline, Week 24
  Absolute change in the percentage of predicted forced expiratory volume in 1 second (%FEV1) from baseline to week 24 of Orkambi®

SECONDARY OUTCOMES:
Z-score of FEV1 | Baseline, Week 24, week 48
  Absolute change in the Z-score of forced expiratory volume in 1 second (FEV1) from baseline to week 24 and to week 48
Percentage of FEV1 | Week 48
  Absolute change in the percentage of predicted forced expiratory volume in 1 second (FEV1) from baseline through week 48
% of FVC | Baseline, Week 24 and week 48
  Absolute change in percent predicted of forced vital capacity (%FVC) from baseline through week 24 and 48
% of RFC | Baseline, Week 24 and week 48
  Absolute change in percent predicted of Functional Residual Capacity (%RFC) from baseline through week 24 and 48
Lung clearance index | Baseline, Week 48
  Absolute change in lung clearance index 2.5 (LCI2.5) from baseline through Week 48
Height | Baseline, Week 24 and week 48
  Absolute change in height-for-age-z-score from baseline to week 24 and 48
Weight | Baseline, Week 24 and week 48
  Absolute change in weight-for-age-z-score from baseline to week 24 and 48
colony forming unit (CFU) | Baseline, Week 24 and week 48
  Absolute change in colony forming unit (CFU) of sputum microorganisms from baseline to week 24 and 48
Number of exacerbations | Baseline, Week 48
  Number of exacerbations to week 48 in comparison to the year previous treatment with Orkambi®
Sweat Cl- | Baseline, Week 48
  Absolute change in sweat Cl- from baseline to week 48
Level in Forskolin/IBMXdependant Short Circuit Current | Baseline
  Level in Forskolin/IBMXdependant Short Circuit Current change in patient nasal epithelial (HNE) cells incubated with Lumacaftor/Ivacaftor
percentage of cells displaying apical staining | baseline
  Correction of CFTR expression at the apical membrane in HNE cells incubated with Lumacaftor/Ivacaftor, assessed by the percentage of cells displaying apical staining.
Area under the curve (AUC) of Lumacaftor/Ivacaftor | Week 24, week 48
  Pharmacokinetic parameters of Lumacaftor, M28-lumacaftor, Ivacaftor, M1-ivacaftor, and M6-ivacaftor
Drug concentrations of Lumacaftor/Ivacaftor | Week 24, week 48
  Pharmacokinetic parameters of Lumacaftor, M28-lumacaftor, Ivacaftor, M1-ivacaftor, and M6-ivacaftor

CONTACTS AND LOCATIONS:
Overall Officials: ISABELLE SERMET, PhD, Principal Investigator — Hospital Necker Enfants Malades
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Bouazza N, Urien S, Foissac F, Choupeaux L, Lui G, Froelicher Bournaud L, Rouillon S, Zheng Y, Bardin E, Stremler N, Bessaci K, Bihouee T, Coirier-Duet E, Marguet C, Deneuville E, Laurans M, Reix P, Gerardin M, Mittaine M, Epaud R, Thumerelle C, Weiss L, Berthaud R, Semeraro M, Treluyer JM, Benaboud S, Sermet-Gaudelus I. Lumacaftor/Ivacaftor Population Pharmacokinetics in Pediatric Patients with Cystic Fibrosis: A First Step Toward Personalized Therapy. Clin Pharmacokinet. 2024 Mar;63(3):333-342. doi: 10.1007/s40262-023-01342-3. Epub 2024 Feb 4. PMID 38310629